CLINICAL TRIAL: NCT05587855
Title: Effects of eCulinary Medicine Emphasizing Herbs and Spices to Increase Vegetable Consumption Among Adults With Hypertension
Brief Title: eCulinary Medicine Emphasizing Herbs/Spices to Increase Vegetable Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: McCormick and Company, Inc. (Industry)
Responsible Party: Principal Investigator, Shannon Galyean, Assistant Professor/Registered Dietitian Nutritionist, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2021-446
Record Dates: First submitted 2022-09-16; First posted 2022-10-20 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Hypertension; Diet, Healthy; Culinary Medicine
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This will be a 6-week randomized controlled intervention. Participants with hypertension will be assigned to an eCulinary medicine group (E-group) or control that will receive recipes without the eCulinary intervention (C-group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eCulinary Medicine Group (E-group) (Experimental): The intervention group will receive weekly cooking demonstrations and education videos via electronic links to use herbs and spices to increase vegetables and reduce sodium in the diet over six weeks
  Interventions: Other: E-group
- Control Group (C-group) (No Intervention): The control group participants will receive usual care from their physician's clinic and the recipes but without the eCulinary intervention over 6 weeks.

INTERVENTIONS:
Other: E-group — Participants with Hypertension will be assigned to eCulinary medicine
  Arms: eCulinary Medicine Group (E-group)

SUMMARY:
e-Culinary medicine emphasizes on herbs and spices, will increase consumption of vegetables and reduce sodium in the diets of people with hypertension and lead to a more favorable health profile.

DETAILED DESCRIPTION:
This will be a randomized controlled intervention in collaboration with physician care clinics. Participants with hypertension will be assigned to an eCulinary medicine group (E-group) or control that will receive recipes without the eCulinary intervention (C-group). The intervention group will receive weekly cooking demonstration videos, a one-time nutrition education session based on the content of the Nutrition Care Manual from the Academy of Nutrition and Dietetics, a bi-weekly phone visit, and will be given a digital blood pressure monitor and a digital weight scale. The cooking demonstrations will focus on utilizing herbs and spices in the preparation of various vegetables using different cooking methods aimed to reduce sodium and increase vegetable consumption. The control group will receive only recipes from the eCulinary intervention as well digital blood pressure monitor and a digital weight scale.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis hypertension
* Age above 18

Exclusion Criteria:

* Use of tobacco
* Self-reported history of chronic diseases other than hypertension
* Allergy to any food
* Pregnant or lactating
* Alcohol or drug dependence

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Dietary Intake | at baseline
  Dietary intake by National Cancer Institute Dietary Screener Questionnaire included a section with questions about 27 individual culinary herbs and spices. Scale is A-K and we use this to compare pre and post intervention for higher intakes of vegetables.
Dietary Intake | 6 weeks
  Dietary intake by National Cancer Institute Dietary Screener Questionnaire included a section with questions about 27 individual culinary herbs and spices. Scale is A-K and we use this to compare pre and post intervention for higher intakes of vegetables.
Dietary Intake | 1 month post intervention
  Dietary intake by National Cancer Institute Dietary Screener Questionnaire included a section with questions about 27 individual culinary herbs and spices. Scale is A-K and we use this to compare pre and post intervention for higher intakes of vegetables.
Diet Quality | at baseline
  Diet quality using the Healthy Eating Index (HEI), a standardized scoring metric that can be used to score any set of foods to evaluate quality as compared to the Dietary Guidelines for Americans. The scores range from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Americans.
Diet Quality | 2 weeks
  Diet quality using the Healthy Eating Index (HEI), a standardized scoring metric that can be used to score any set of foods to evaluate quality as compared to the Dietary Guidelines for Americans. The scores range from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Americans.
Diet Quality | 4 weeks
  Diet quality using the Healthy Eating Index (HEI), a standardized scoring metric that can be used to score any set of foods to evaluate quality as compared to the Dietary Guidelines for Americans. The scores range from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Americans.
Diet Quality | 6 weeks
  Diet quality using the Healthy Eating Index (HEI), a standardized scoring metric that can be used to score any set of foods to evaluate quality as compared to the Dietary Guidelines for Americans. The scores range from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Americans.
Diet Quality | 1 month post intervention
  Diet quality using the Healthy Eating Index (HEI), a standardized scoring metric that can be used to score any set of foods to evaluate quality as compared to the Dietary Guidelines for Americans. The scores range from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Americans.
Cooking effectiveness evaluation | 2 weeks
  A quantitative and qualitative evaluation of the eCulinary program, using a pre-test/post-test study and cooking effectiveness over time. The test asks questions regarding the recipes that were used, number of times a recipe was used, and if it was useful.
Cooking effectiveness evaluation | 4 weeks
  A quantitative and qualitative evaluation of the eCulinary program, using a pre-test/post-test study and cooking effectiveness over time. The test asks questions regarding the recipes that were used, number of times a recipe was used, and if it was useful.
Cooking effectiveness evaluation | 6 weeks
  A quantitative and qualitative evaluation of the eCulinary program, using a pre-test/post-test study and cooking effectiveness over time. The test asks questions regarding the recipes that were used, number of times a recipe was used, and if it was useful.
Cooking effectiveness evaluation | 1 month post intervention
  A quantitative and qualitative evaluation of the eCulinary program, using a pre-test/post-test study and cooking effectiveness over time. The test asks questions regarding the recipes that were used, number of times a recipe was used, and if it was useful.

SECONDARY OUTCOMES:
Systolic or Diastolic Blood Pressure | at baseline
  Participants will receive an Omron 3 Series Upper Arm Blood Pressure Monitor (HBPM) (Model BP7100). They will be instructed to use their device to take readings to track over time and share with the researchers and health care providers.
Systolic or Diastolic Blood Pressure | 2 weeks
  Participants will receive an Omron 3 Series Upper Arm Blood Pressure Monitor (HBPM) (Model BP7100). They will be instructed to use their device to take readings to track over time and share with the researchers and health care providers.
Systolic or Diastolic Blood Pressure | 4 weeks
  Participants will receive an Omron 3 Series Upper Arm Blood Pressure Monitor (HBPM) (Model BP7100). They will be instructed to use their device to take readings to track over time and share with the researchers and health care providers.
Systolic or Diastolic Blood Pressure | 6 weeks
  Participants will receive an Omron 3 Series Upper Arm Blood Pressure Monitor (HBPM) (Model BP7100). They will be instructed to use their device to take readings to track over time and share with the researchers and health care providers.
Systolic or Diastolic Blood Pressure | 1 month post intervention
  Participants will receive an Omron 3 Series Upper Arm Blood Pressure Monitor (HBPM) (Model BP7100). They will be instructed to use their device to take readings to track over time and share with the researchers and health care providers.
Body Weight | at baseline
  Participants will receive a Doran DS500 Digital Flat Floor Scale, instructions about using their device for home weight monitoring. They will be instructed to use their device to take readings to track over time and share with the researchers and health care providers.
Body Weight | 2 weeks
  Participants will receive a Doran DS500 Digital Flat Floor Scale, instructions about using their device for home weight monitoring. They will be instructed to use their device to take readings to track over time and share with the researchers and health care providers.
Body Weight | 4 weeks
  Participants will receive a Doran DS500 Digital Flat Floor Scale, instructions about using their device for home weight monitoring. They will be instructed to use their device to take readings to track over time and share with the researchers and health care providers.
Body Weight | 6 weeks
  Participants will receive a Doran DS500 Digital Flat Floor Scale, instructions about using their device for home weight monitoring. They will be instructed to use their device to take readings to track over time and share with the researchers and health care providers.
Body Weight | 1 month post intervention
  Participants will receive a Doran DS500 Digital Flat Floor Scale, instructions about using their device for home weight monitoring. They will be instructed to use their device to take readings to track over time and share with the researchers and health care providers.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Galyean, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] (CDC) CfDCaP. Hypertension Cascade: Hypertension Prevalence, Treatment and Control Estimates Among US Adults Aged 18 Years and Older Applying the Criteria From the American College of Cardiology and American Heart Association's 2017 Hypertension Guideline-NHANES 2013-2016 2019 [cited 2021]. Available from: Million Hearts® (hhs.gov).
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):1269-1324. doi: 10.1161/HYP.0000000000000066. Epub 2017 Nov 13. No abstract available. PMID 29133354
- [Background] Aburto NJ, Ziolkovska A, Hooper L, Elliott P, Cappuccio FP, Meerpohl JJ. Effect of lower sodium intake on health: systematic review and meta-analyses. BMJ. 2013 Apr 3;346:f1326. doi: 10.1136/bmj.f1326. PMID 23558163
- [Background] Bibbins-Domingo K, Chertow GM, Coxson PG, Moran A, Lightwood JM, Pletcher MJ, Goldman L. Projected effect of dietary salt reductions on future cardiovascular disease. N Engl J Med. 2010 Feb 18;362(7):590-9. doi: 10.1056/NEJMoa0907355. Epub 2010 Jan 20. PMID 20089957
- [Background] Palar K, Sturm R. Potential societal savings from reduced sodium consumption in the U.S. adult population. Am J Health Promot. 2009 Sep-Oct;24(1):49-57. doi: 10.4278/ajhp.080826-QUAN-164. PMID 19750962
- [Background] Fritts JR, Fort C, Quinn Corr A, Liang Q, Alla L, Cravener T, et al. Herbs and spices increase liking and preference for vegetables among rural high school students. Food Quality and Preference. 2018;68:125-34. doi: https://doi.org/10.1016/j.foodqual.2018.02.013.
- [Background] Anderson CA, Cobb LK, Miller ER 3rd, Woodward M, Hottenstein A, Chang AR, Mongraw-Chaffin M, White K, Charleston J, Tanaka T, Thomas L, Appel LJ. Effects of a behavioral intervention that emphasizes spices and herbs on adherence to recommended sodium intake: results of the SPICE randomized clinical trial. Am J Clin Nutr. 2015 Sep;102(3):671-9. doi: 10.3945/ajcn.114.100750. Epub 2015 Aug 12. PMID 26269371
- [Background] Wang C, Lee Y, Lee SY. Consumer acceptance of model soup system with varying levels of herbs and salt. J Food Sci. 2014 Oct;79(10):S2098-106. doi: 10.1111/1750-3841.12637. Epub 2014 Sep 12. PMID 25220863
- [Background] Ghawi SK, Rowland I, Methven L. Enhancing consumer liking of low salt tomato soup over repeated exposure by herb and spice seasonings. Appetite. 2014 Oct;81:20-9. doi: 10.1016/j.appet.2014.05.029. Epub 2014 May 28. PMID 24879887
- [Background] Aburto NJ, Hanson S, Gutierrez H, Hooper L, Elliott P, Cappuccio FP. Effect of increased potassium intake on cardiovascular risk factors and disease: systematic review and meta-analyses. BMJ. 2013 Apr 3;346:f1378. doi: 10.1136/bmj.f1378. PMID 23558164
- [Background] Services USDoAaUSDoHaH. Dietary Guidelines for Americans, 2020-2025 2020 [cited 2021].
- [Background] Kimmons J, Gillespie C, Seymour J, Serdula M, Blanck HM. Fruit and vegetable intake among adolescents and adults in the United States: percentage meeting individualized recommendations. Medscape J Med. 2009;11(1):26. Epub 2009 Jan 26. PMID 19295947
- [Background] Lucan SC, Barg FK, Long JA. Promoters and barriers to fruit, vegetable, and fast-food consumption among urban, low-income African Americans--a qualitative approach. Am J Public Health. 2010 Apr;100(4):631-5. doi: 10.2105/AJPH.2009.172692. Epub 2010 Feb 18. PMID 20167885
- [Background] Irl B H, Evert A, Fleming A, Gaudiani LM, Guggenmos KJ, Kaufer DI, McGill JB, Verderese CA, Martinez J. Culinary Medicine: Advancing a Framework for Healthier Eating to Improve Chronic Disease Management and Prevention. Clin Ther. 2019 Oct;41(10):2184-2198. doi: 10.1016/j.clinthera.2019.08.009. Epub 2019 Sep 20. PMID 31543284
- [Background] Casagrande SS, Gary-Webb TL. Chapter 8 - Trends in US Adult Fruit and Vegetable Consumption. In: Watson RR, Preedy VR, editors. Bioactive Foods in Promoting Health. San Diego: Academic Press; 2010. p. 111-30.
- [Background] Kalantar-Zadeh K, Mattix-Kramer HJ, Moore LW. Culinary Medicine as a Core Component of the Medical Nutrition Therapy for Kidney Health and Disease. J Ren Nutr. 2021 Jan;31(1):1-4. doi: 10.1053/j.jrn.2020.11.002. No abstract available. PMID 33357519
- [Background] Brors G, Pettersen TR, Hansen TB, Fridlund B, Holvold LB, Lund H, Norekval TM. Modes of e-Health delivery in secondary prevention programmes for patients with coronary artery disease: a systematic review. BMC Health Serv Res. 2019 Jun 10;19(1):364. doi: 10.1186/s12913-019-4106-1. PMID 31182100